CLINICAL TRIAL: NCT02835898
Title: The Effect of Periodontal Therapy on Epigenetic Changes: A Pilot Study
Brief Title: Epigenetics and Periodontal Treatment
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Giulio Rasperini, Professor of periodontology, University of Milan
Other Study IDs: Epigenetics
Record Dates: First submitted 2016-07-07; First posted 2016-07-18 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gingival biopsies will be collected in tubes that contain Allprotect tissue reagent (100 ml, Qiagen, USA), to immediately and effectively stabilize the DNA in tissues, based on the manufacturer's instructions. Tubes containing the reagent will be stored at 2-8 C. Later DNA/RNA will be purified using AllPrep DNA/RNA Mini Kit (50 ml, Qiagen, USA), following the manufacturer's instructions. With this approach, quantitative gene expression of specific cytokines is possible.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Test Group: Patients with periodontal disease that need conventional periodontal treatment
  Interventions: Other: Conventional periodontal treatment
- Control Group: Periodontally-healthy individuals.

INTERVENTIONS:
Other: Conventional periodontal treatment — Conventional routine periodontal treatment will be done for patients in test group
  Groups: Test Group

SUMMARY:
Objective: The aim of this pilot study is to evaluate the alterations of epigenetic patterns in periodontally diseased individuals, before and after periodontal treatment, also in comparison to periodontally healthy patients.

Materials & methods: Twenty patients were voluntarily enrolled in two groups: 10 participants with healthy periodontium, and 10 participants with chronic periodontitis. Clinical parameters were recorded and gingival biopsies were collected within the following timelines: At baseline (for both groups), after 15 days (for the diseased group only) and after two months (for the diseased group only).

DETAILED DESCRIPTION:
Study Design Baseline: Before harvesting gingival biopsies, bleeding on probing (BOP), periodontal pocket depth (PPD) and clinical attachment level (CAL) were registered at the biopsy site, for all study participants. Following the registration of the clinical parameters, gingival biopsies were obtained from the periodontally-healthy individuals during crown lengthening surgery or surgical removal of wisdom teeth. In the periodontally-diseased group, biopsies were harvested from two sites: healthy site and periodontally-involved site. After harvesting of biopsies, patients with periodontal disease underwent scaling and root planing.

Two weeks after periodontal treatment: Clinical parameters were registered and gingival biopsies were harvested (from two sites) for the periodontally-diseased group only, to evaluate if the epigenetic patterns (DNA methylation) were altered by conventional periodontal therapy, in comparison to the patterns observed at baseline for both diseased and healthy groups.

Two months after initial periodontal treatment: Clinical parameters were registered and gingival biopsies were harvested (from two sites) for the periodontally-diseased group only, to evaluate if the epigenetic patterns were still altered by conventional periodontal therapy, in comparison to the patterns observed at baseline for both diseased and healthy groups, and at 15 days for the diseased group.

ELIGIBILITY:
Inclusion Criteria:

* All participants should be systemically healthy
* All patients should be non-smokers
* Study participants should not be on antibiotics or non-steroidal anti-inflammatory drugs (NSAIDs) within one month before enrolment in the study
* All participants should be of a Caucasian ethnicity

Exclusion Criteria:

* Patients with systemic diseases
* Smoking patients
* Patients taking antibiotics or NSAIDs

Ages: 26 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups: ten patients with chronic periodontitis and ten individuals with healthy periodontium
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Changes in in the levels of DNA methylation (type of epigenetic modification) following periodontal therapy | 0, 15 days after periodontal therapy, 2 months after periodontal therapy

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Rasperini, DDS, Principal Investigator — University of Milan
Locations (1):
- Studio Odontoiatrico Professor Rasperini, Piacenza, PC, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Asa'ad F, Bollati V, Pagni G, Castilho RM, Rossi E, Pomingi F, Tarantini L, Consonni D, Giannobile WV, Rasperini G. Evaluation of DNA methylation of inflammatory genes following treatment of chronic periodontitis: A pilot case-control study. J Clin Periodontol. 2017 Sep;44(9):905-914. doi: 10.1111/jcpe.12783. Epub 2017 Aug 17. PMID 28736819